# National Longitudinal Cohort of Hematological Diseases -Acute Myeloid Leukemia (NICHE-AML)

Applicant: Institute of Hematology & Blood Diseases Hospital

Version: 1.0

Date: 30-Jul-2020

National Longitudinal Cohort of Hematological Diseases-Acute Myeloid Leukemia (NICHE-AML)

## Background

Hematological diseases are disorders of the blood and hematopoietic organs. The current hematological cohorts are mostly based on single-center or multi-center cases, or cohorts with limited sample size in China. There is a lack of comprehensive and large-scale prospective cohort studies in hematology.

## Objectives

The objectives of this study is to investigate the incidence and risk factors of AML, and to analyze the treatment methods, prognosis and medical expenses of these patients in China.

# Subjects

Patients who were diagnosed with AML in the investigating hospitals from January 1, 2020.

### Method

The NICHE-AML will collect basic information, diagnostic and treatment information, as well as medical expense information of patients from medical records. The study will use questionnaire to measure the exposure of patients, and prospectively follow-up to collect the prognosis information.